CLINICAL TRIAL: NCT01700478
Title: A Trial Comparing The Use Of Rectal Plus Perivascular Vasopressin With Perivascular Vasopressin Alone To Decrease Bleeding At The Time Of Myomectomy
Brief Title: Study of the Use of Misoprostol to Decrease Bleeding During a Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of the West Indies (Other)
Responsible Party: Principal Investigator, Dr Sharifa Frederick, Doctor, University Hospital of the West Indies
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: MV-001
Record Dates: First submitted 2012-09-25; First posted 2012-10-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2012-10

CONDITIONS: Hemorrhage
Keywords: Myomectomy
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Misoprostol + vasopressin, Vasopressin (Experimental): Misoprostol 400ug given rectally one hour before surgery.
  Interventions: Drug: Misoprostol + vasopressin; Drug: Vasopressin

INTERVENTIONS:
Drug: Misoprostol + vasopressin — 400ug of misoprostol is given per rectum, one hour prior to surgery. Vasopressin is used at the time of surgery.
  Other Names: Cytotec
Drug: Vasopressin — Vasopressin was used in all patients during surgery.
  Other Names: Anti-diuretic hormone

SUMMARY:
This study was done to determine if the use of a combination of preoperative rectal misoprostol 400µg used with intraoperative perivascular vasopressin is better than perivascular vasopressin used alone to decrease bleeding at myomectomy.

DETAILED DESCRIPTION:
A myomectomy is a fertility sparing procedure in which fibroids are removed from the uterus. This procedure can be associated with significant blood loss which can result in significant morbidity and mortality. The drug misoprostol which has been been use in the treatment of postpartum hemorrhage was given to subset of patients who were scheduled to undergo elective myomectomy at the University hospital of the West Indies and from the private practice of the participating doctors who were invited to participate in the study. Patients were randomized to receive or not to receive pre-operative rectal misoprostol 400µg, 60 minutes before surgery. Twenty five patients received misoprostol and twenty patients did not.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic fibroids who desire future fertility and or who wish to maintain their uterus.

Exclusion Criteria:

* patients who have had previous myomectomy or previous pelvic surgery.
* patients who are severely anemic or who have significant medical conditions such as cardiac or pulmonary disease.
* patients who refuse to participate or give consent to the procedures. Patients with a known allergy to any of the study drugs.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Blood loss in millilitres | At the time of surgery

SECONDARY OUTCOMES:
A change in hemoglobin grams per decilitre | At baseline and 24hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sharifa K Frederick, dM, Principal Investigator — University Hospital of the West Indies
Locations (1):
- University Hospital of the West Indies, Kingston, Jamaica

REFERENCES:
- [Derived] Frederick S, Frederick J, Fletcher H, Reid M, Hardie M, Gardner W. A trial comparing the use of rectal misoprostol plus perivascular vasopressin with perivascular vasopressin alone to decrease myometrial bleeding at the time of abdominal myomectomy. Fertil Steril. 2013 Oct;100(4):1044-9. doi: 10.1016/j.fertnstert.2013.06.022. Epub 2013 Jul 19. PMID 23876539